CLINICAL TRIAL: NCT06876857
Title: University of Central Florida CereBank
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00007544
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Biospecimen Donation; Brain Injury; Brain Diseases
Keywords: donate; biobank; brain; biospecimen; Alzheimer's Disease; Autism; Huntington's Disease
MeSH Terms: conditions — Brain Injuries; Brain Diseases; Alzheimer Disease; Autistic Disorder; Huntington Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Donated brain tissue and biospecimens: Persons with brain disease and/ or brain trauma to be used to support research studies aimed at improving the diagnosis and treatment of brain diseases.

SUMMARY:
Millions of persons are affected by brain diseases. The CereBank will be used to support research studies aimed at improving the diagnosis and treatment of brain diseases. Brain diseases can be inherited; developed due to diseases or aging; or can be due to trauma. The Central Florida does not have a brain biobank to meet the needs of research. Therefore, it is necessary for the University of Central Florida to establish a brain biobank.

DETAILED DESCRIPTION:
The purpose of the University of Central CereBank is to be a brain repository to support the research of the faculty of the University of Central Florida College of Medicine. These research studies aim at improving the diagnosis and treatment of brain diseases, such as dementia, to advance medicine. The donated brains will be used for research and educational purposes.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older.
* Able to provide informed consent. Persons who are unable to provide an informed consent will need a Legally Authorized Representative (LAR) to sign the informed consent.

Exclusion Criteria:

* minors (under age 18).
* prisoners.
* pregnant women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will donate brain tissue for research and education, aimed at improving the diagnosis and treatment of brain diseases.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2075-02-25 (Estimated); Study Completion 2075-02-25 (Estimated)

PRIMARY OUTCOMES:
Receipt of donated brain tissue and biospecimens for research and educational purposes | 75 years
  The UCF CereBank will be used to support research studies aimed at improving the diagnosis and treatment of brain diseases. Brain diseases can be inherited; developed due to diseases or aging; or can be due to trauma.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States